CLINICAL TRIAL: NCT01896323
Title: An Open-Label, Two-Period, Fixed-Sequence Study to Evaluate the Effect of Multiple Doses of Ketoconazole on the Single Dose Pharmacokinetics of CC-223 in Healthy Adult Male Subjects
Brief Title: CC-223 and Ketoconazole Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CC-223-CP-003
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — CC-223; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC-223 (Experimental): CC-223 administration on study day 1 of Period 1 and study day 5 of Period 2
  Interventions: Drug: CC-223
- Ketokonazole (Active Comparator): Ketoconazole administration on study days 1 through 8 of Period 2
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: CC-223 — CC-223 20 mg tablets
  Arms: CC-223
Drug: Ketoconazole — Ketoconazole 400 mg tablets
  Other Names: Nizoral
  Arms: Ketokonazole

SUMMARY:
This is a single-center open-label study to compare how CC-223 (the study drug being investigated) interacts with the drug ketoconazole.

DETAILED DESCRIPTION:
This is a 2 period study, which lasts about 6 weeks long. About 14 males will be entered into the study, during which they will receive the study drug (a single dose of 20 mg CC-223) 400 mg ketoconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign a written informed consent form before participation.
2. Must be able to communicate with the study doctor, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Healthy male subject of any race between 18 to 65 years of age, and in good health as determined by a physical examination.

   - For males: Agree to use barrier contraception not made of natural (animal) membrane (for example, latex or polyurethane condoms are acceptable) when engaging in sexual activity with a female of child-bearing potential while on study medication, and for at least 28 days after the last dose of study medication.
4. Must have a body mass index between 18 and 33 kilograms/meter squared.
5. Clinical laboratory tests must be within normal limits or acceptable to the study doctor.
6. Must not have a fever, with a blood pressure between 90/50 to 140/90 millimeters of mercury, and pulse rate: between 40 to 110 beats per minute.
7. Must have a normal or clinically acceptable 12-lead electrocardiogram.

Exclusion Criteria:

1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.
2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
3. Used any prescribed or topical medication within one month before the first dose of study drug, unless consultation between the sponsor and the study doctor.
4. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 2 weeks (30 days for St. John's Wort®) of the first dose administration, unless sponsor agreement is obtained.
5. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion of the study drug, for example, bariatric procedure.
6. Donated blood or plasma within 2 months before the first dose of study drug.
7. History of drug abuse within 2 years before dosing, or a positive drug screening test reflecting consumption of illicit drugs.
8. History of alcohol abuse within 2 years before dosing, or positive alcohol screen.
9. Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen, or hepatitis C antibody, or have a positive result to the test for Human Immune virus antibodies at Screening.
10. Exposed to an investigational drug within one month 30 days before the first dose of study drug.
11. Smoke more than 10 cigarettes per day, or the equivalent in other tobacco products.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2013-08-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | up to 96 hours post dose
  AUC-area under the plasma concentration-time curve;
Pharmacokinetics | up to 96 hours post dose
  Cmax-maximum observed plasma concentration
Pharmacokinetics | up to 96 hours post dose
  Tmax - Time to maximum observed plasma concentration
Pharmacokinetics | up to 96 hours post dose
  t½ - terminal elimination half-life in plasma

SECONDARY OUTCOMES:
Adverse Events | Up to 28 days after last dose of study drug
  Number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation

REFERENCES:
- [Background] Tong Z, Narayanan R, Atsriku C, Nissel J, Li Y, Liu H, Wang X, Surapaneni S. Assessment of drug-drug interaction potential and PBPK modeling of CC-223, a potent inhibitor of the mammalian target of rapamycin kinase. Xenobiotica. 2019 Jan;49(1):54-70. doi: 10.1080/00498254.2018.1424377. Epub 2018 Jan 17. PMID 29297772